CLINICAL TRIAL: NCT03408717
Title: Evaluation And Risk Assessment For Persistent Postsurgical Pain After Breast Surgery: A Prospective Cohort Study (Breast CAncer Surgery Postsurgical Pain)
Brief Title: Evaluation And Risk Assessment For Persistent Postsurgical Pain After Breast Surgery
Acronym: B-CAPP
Status: Active, not recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/2805
Record Dates: First submitted 2017-12-28; First posted 2018-01-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Chronic Pain; Acute Pain; Depression, Anxiety
Keywords: Breast cancer; Chronic pain; Acute Pain; Depression; Anxiety
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Acute Pain; Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from venous blood using the Puregene method at the Research Laboratory of the mentioned site. Known functional polymorphisms in Catechol-O-methyltransferase (COMT), Calcium channel, voltage-dependent, gamma subunit (CACNG2) and Sodium Voltage-Gated Channel Alpha Subunit 9 (SCN9A) gene with evidence of associations with depression, pain, stress and anxiety would be determined by the Taqman allelic discrimination assay method. Alleles will be called using the software. Genetic data will be analyzed for association with the presence of persistent pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persistent post surgical pain (PPSP): Questionnaires, Mechanical Temporal Summation assessment and pain threshold assessment will be assigned to patient. Within this cohort, some patients will have high pain score recorded (persistent pain) during the follow-up evaluations at 4 and 6 months.
  Interventions: Other: Questionnaires; Other: Mechanical Temporal Summation assessment; Other: Pain threshold assessment

INTERVENTIONS:
Other: Questionnaires — Questionnaires including Pain catastrophizing scale (PCS), Central Sensitisation Inventory (CSI), Coping Strategies Questionnaire-Revised (CSQ-R), Brief Symptom Inventory-18 (BSI-18), Perceived Stress Scale (PSS), EQ-5D-3L and Eysenck Personality Questionnaire (EPQ) will be administered to the patient.
Other: Mechanical Temporal Summation assessment — A 180 gram von Frey filament is applied on the subject's forearm. Patient will then be asked to rate the pinprick pain score on a verbal rating scale, 0-100. Following this, 10 consecutive touches at random locations are applied with a 1 second interstimulus interval and within a 1 cm diameter circle. The patient will then be asked to rate the 10th pain score (0-100). The Mechanical Temporal Summation Score is obtained by the difference between the 11th pain score and the 1st pain score. If the score is greater than zero, the patient is implied to have presence of Mechanical Temporal Summation.
  Other Names: MTS
Other: Pain threshold assessment — Pressure is applied 90 degree straight down force on the subject's right/left centre of the trapezius muscle using an algometer, with a speed of pressure ~ 1kgf/s. The above procedure is then repeated 3 times at each site (left/right) which is indicated on the pressure mark with each time having the reading recorded. When patient shows no response ≥ 6kgf, the threshold is recorded as 6kgf. The patient upon feeling pain will say stop or raise the hand to terminate the test. The mean value is obtained by averaging the readings and will then be recorded as the threshold estimate.
  Other Names: Pressure pain

SUMMARY:
Pre-existing pain and severe postoperative pain are predictors of persistent pain after surgery, but a complete understanding on the development of persistent pain is still lacking. The study aims to identify clinically relevant and genetic risk factors for persistent postsurgical pain that can be reliably distinguished statistically.

DETAILED DESCRIPTION:
The study will focus on: (i) risk factors representing biopsychosocial processes that influence chronic pain, such as pain and psychological vulnerability; (ii) genetic factors relating to mechanistic pathways to persistent pain generation. Patients will be recruited from those undergoing breast cancer surgery at the mentioned site. Pain and anxiety assessment will be conducted via visual analogue scoring, mechanical temporal summation assessment and a series of questionnaires. After the surgery, all patients will be given appropriate analgesia, and the pain score and analgesia usage will be recorded. Phone survey will be conducted 4 and 6 months, respectively, after surgery to determine the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 - 80 year old;
* Healthy and/or have systemic medical conditions as reviewed by anaesthetist for surgery (ASA 1-3);
* Undergoing breast cancer surgery.

Exclusion Criteria:

* History of intravenous drug or opioid abuse;
* Current chronic daily treatment with corticosteroids (excluding inhaled steroids);
* Previous history of chronic pain syndrome;
* Obstetric patients.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females who undergo breast surgery will be included in this study.
Study Population: Patients undergoing breast cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Persistent pain at 4 months after surgery | 4 months after surgery
  Persistent pain is defined as having one of the below criteria at 4 months after surgery:
  i) having pain score at rest (Numeric Rating Scale 0 to 100) of 30 or more; or ii) having pain score on movement (Numeric Rating Scale 0 to 100) of 30 or more; or iii) or "yes" to one of the seven questions on the presence of pain in daily life activities (mood, walking, carrying heavy loads, work, relations with people, sleep, enjoyment of life)

SECONDARY OUTCOMES:
Persistent pain at 6 months after surgery | 6 months after surgery
  Persistent pain is defined as having one of the below criteria at 4 months after surgery:
  i) having pain score at rest (Numeric Rating Scale 0 to 100) of 30 or more; or ii) having pain score on movement (Numeric Rating Scale 0 to 100) of 30 or more; or iii) or "yes" to one of the seven questions on the presence of pain in daily life activities (mood, walking, carrying heavy loads, work, relations with people, sleep, enjoyment of life)
Maximum Acute post-operative pain score | Up to 3 days after surgery
  The maximum number of patient-reported post-operative pain score (Numeric Rating Scale 0 to 100) at 0 - 72 hours
Opioid consumption | Up to 3 days after surgery
  The total opioid consumption (morphine/ fentanyl/ hydromorphone/ oxycodone/ hydrocodone etc) throughout the 72 hours. The opioid consumption will be converted using oral morphine equivalent (OME) conversion calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital; Ashraf Habib, MBBCh, FRCA, Principal Investigator — Duke University
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03408717/Prot_SAP_000.pdf